CLINICAL TRIAL: NCT05758363
Title: Randomized Clinical Trial to Evaluate the Efficacy of a Dietary Supplement on Weight Loss and Psychological Wellbeing in Overweight Individuals
Brief Title: Effect of a Dietary Supplement on Weight Loss and Psychological Wellbeing in Overweight Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Desirée Victoria Montesinos, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE012309
Record Dates: First submitted 2023-02-20; First posted 2023-03-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Dietary Supplements; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Consumption of dietary supplement capsules for 6 months.
  Interventions: Dietary Supplement: Consumption of dietary supplement.
- Control Group (Placebo Comparator): Identically appearing placebo capsules consumed for 6 months.
  Interventions: Other: Consumption of control product

INTERVENTIONS:
Dietary Supplement: Consumption of dietary supplement. — Consumption of a dietary supplement rich in glutathione, selenium, zinc, vitamin D and EPA/DHA. 1 capsule per day of the dietary supplement with breakfast.
  Arms: Experimental Group
Other: Consumption of control product — Consumption of 1 capsule per day of control product of identical appearance with breakfast.
  Arms: Control Group

SUMMARY:
The aim of this randomized, parallel, two-arm, placebo-controlled, double-blind, multicenter clinical trial is to evaluate the efficacy of a dietary supplement on weight loss and psychological well-being in overweight individuals.

DETAILED DESCRIPTION:
The duration of the study will be 6 months during which the investigational product or placebo will be consumed according to the assignment.

Subjects will be randomized to each of the study arms (consumption of the experimental product or control product).

ELIGIBILITY:
Inclusion Criteria:

* Adults (age: 30 - 70 YO)
* BMI over 25 kg/m2.
* Subjects who are smokers or non-smokers, but in any case who do not modify their nicotinic habits during their participation in the study.

Exclusion Criteria:

* Subjects with eating disorders.
* BMI less than 25 Kg/m2.
* History of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Participation in another clinical trial in the three months prior to the study.
* Unwillingness or inability to comply with clinical trial procedures.
* Pregnant woman.
* Participants with an active daily exercise activity.
* Subjects whose condition makes them ineligible for the study at the investigator's discretion.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of weight loss | From baseline to 6 months later
  Evaluation of weight loss by assessment of anthropometric measurements - Waist/hip ratio - Waist/height ratio.

SECONDARY OUTCOMES:
Quality of life by WHOQOL-BREF | From baseline to 6 months later
  World Health Organization Quality of Life Brief version test. The raw scores are transformed into a normalized scale ranging from 4 to 20 and from 0 to 100. Higher scores indicating better quality of life.
Quality of life by SF-36 | From baseline to 6 months later
  Short Form 36 Health Survey Questionnaire (SF-36). The SF-36 contains 36 items that measure eight dimensions or scales. The scores for each dimension will be calculated in both raw and transformed form as indicated in the manual, with higher scores indicating better health status for that particular dimension.
Depression | From baseline to 6 months later
  Beck Depression Inventory test. The score ranges from 0 to 63, where the higher the score, the greater the signs of depression.
Stress | From baseline to 6 months later
  Perceived Stress Scale (PSS). Total scores range from 0 to 56 (higher scores indicate higher levels of stress).
Anxiety | From baseline to 6 months later
  State-Trait Anxiety Inventory (STAI) Test. Scores can vary between 0 to a maximum of 60. Higher scores correlate positively with higher levels of anxiety.
Dietary intake | From baseline to 6 months later
  Registration and subsequent nutritional evaluation with 3-day food frequency questionnaire (FFQ).

CONTACTS AND LOCATIONS:
Locations (1):
- UCAM San Antonio Catholic University of Murcia, Murcia, Spain